CLINICAL TRIAL: NCT05022433
Title: Comparison of the Shukla and UN-1 Formulae in the Placement of the Umbilical Venous Catheter Among Neonates: A Randomized Clinical Study
Brief Title: Comparison of the Shukla and UN-1 Formulae in the Placement of the Umbilical Venous Catheter Among Neonates
Status: Completed | Type: Observational
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-2300
Record Dates: First submitted 2021-08-09; First posted 2021-08-26 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Extreme Prematurity,Extremely Low Birthweight; Extremely Low Birth Weight; Very Low Birth Weight Infant; Neonatal Hypoglycemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Shukla: Shukla is a birth weight based formula to determine the insertional depth of the UVC
  Interventions: Procedure: UVC insertion
- UN-1: UN-1 is a body surface based formula to determine the insertional depth of the UVC
  Interventions: Procedure: UVC insertion

INTERVENTIONS:
Procedure: UVC insertion — To compare two formulae namely UN-1 and Shukla method to estimate the UVC insertion length in achieving optimum UVC tip position.

SUMMARY:
Umbilical vein catheters (UVC) are commonly inserted in newborns especially neonates admitted to the Neonatal Intensive Care Unit (NICU).These catheters are used since 1959. It is a suitable method for parenteral nutrition access and medications administration. Despite the benefits of the UVC, its potential complications must be considered. Thus, it is vital to determine the appropriate penetration length of the UVC.

DETAILED DESCRIPTION:
UVC insertion has benefits and potential complications such as infection, intestinal necrosis, thrombosis, ascites, hydrothorax, cardiac tamponade, cardiac arrhythmias, pleural effusion, pericarditis and pericardial effusion. The complications may be due to insertion of catheter in an inappropriate location. Imaging procedures such as plain thoracoabdominal x-ray is needed after catheter insertion to specify the location of the catheter tip. In addition to preventing complications, insertion of umbilical venous catheter in an appropriate location is essential for umbilical catheterisation effectiveness. There are different methods to determine the length of catheter which must be inserted in umbilical vessels. The UVC formulae are based on either body surface measurement such as Dunn method, Umbilical to Intermammary Distance (UIMD), Umbilical to Nipple Distance (UN)-1 and birthweight based formula method such as Shukla and Modified Shukla. Shukla and UN-1 Methods have been widely used in the world. However, the accuracy of these two methods in estimating the length of umbilical venous catheter has not still demonstrated.

ELIGIBILITY:
Inclusion Criteria:

* All term and preterm newborns requiring UVC insertion will be included in the study.

Exclusion Criteria:

* All neonates with major congenital malformations that interferes with the placement of the UVC will be excluded.

Ages: 0 Days to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All term and preterm newborns admitted in Singapore General Hospital requiring UVC insertion with no major congenital malformation will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2019-06-06 (Actual); Primary Completion 2023-10-11 (Actual); Study Completion 2023-10-11 (Actual)

PRIMARY OUTCOMES:
Comparison of the Shukla and UN-1 formulae in the Placement of the UVC Among Neonates:A Randomized Clinical Study | 14 days
  Using the chest and abdominal X-ray, the distance of the UVC tip position in reference to the diaphragm level is measured.UVC tip position is then labeled as either IDEAL,SHORT or DEEP position. Ideal position is defined as the UVC tip is at the diaphragm level or +/- 0.5cm distance from the diaphragm. Short UVC is defined if the UVC tip is >0.5 cm below the diaphragm.Deep UVC position is defined as if the UVC tip is > 0.5cm above the diaphragm.

SECONDARY OUTCOMES:
Comparison of the Shukla and UN-1 formulae in the Placement of the UVC Among Neonates:A Randomized Clinical Study | 14 days
  Using the chest and abdominal X-ray, the distance of the UVC tip position in reference between the upper border of T9 to the lower border of T10 level is measured. UVC tip position is then labeled as IDEAL, SHORT and DEEP UVC position.Ideal position is defined as the UVC tip position in between the level of the upper border of T9 to the lower border of T10. Short UVC if the tip is below the lower border of T10. Deep UVC position is defined as the UVC tip above the upper border of T9.

CONTACTS AND LOCATIONS:
Overall Officials: MARY GRACE S TAN, MD, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided